CLINICAL TRIAL: NCT06945861
Title: Immunological Aspects of Thrombotic Thrombocytopenic Purpura (TTP): Characterisation of B and T Lymphocytes Specific for the ADAMTS13 Autoantigen and Therapeutic Implications
Brief Title: Immunological Aspect of Thrombotic Thrombocytopenic Purpura (TTP)
Acronym: Lympho-PTT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/308/OB; IDRCB : 2023-A00455-40 (Other: ANSM)
Record Dates: First submitted 2025-04-07; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-05

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP)
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The aim of whole blood sampling is to characterise phenotypically and functionally the ADAMTS13-specific memory B lymphocytes and autoreactive T lymphocytes, in particular follicular helper T lymphocytes, in the acute phase of the disease, but also during its progression after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: patients in the acute phase of TTP: Consultation or hospitalisation when TTP is diagnosed, before treatment is initiated
- Groupe 2 : patient in durable remission with ADAMTS13 activity > 10%.: Follow-up consultation
- Groupe 3 : patient in remission with ADAMTS13 activity < 10%.: Follow-up consultation before initiation of pre-emptive treatment
- Group 4: relapsing patients: Consultation or hospitalisation at the time of relapse, before treatment is initiated

SUMMARY:
The general objective of the proposed project is to characterise phenotypically and functionally ADAMTS13-specific memory B lymphocytes and autoreactive T lymphocytes, in particular follicular helper T lymphocytes, in the acute phase of the disease, but also during its progression after treatment. The aim is to highlight their contribution to the initial pathogenic process, their evolution under treatment, and also their involvement in patients who are refractory to immunosuppressive therapies and during relapses. The aim of this project is to identify early phenotypic or functional parameters that are predictive of relapse and that can be used for personalised optimisation of treatment to maintain remission.

DETAILED DESCRIPTION:
Thrombotic thrombocytopenic purpura (TTP) is characterised by profound thrombocytopenia, haemolytic anaemia and organ dysfunction (cardiac, neurological or renal). The current treatment strategy includes plasma exchange, corticosteroid therapy, rituximab and caplacizumab, a bivalent humanised 'nanobody' targeting the A1 domain of factor Willebrand, thereby inhibiting platelet adhesion. Several response profiles to this first line of treatment have been observed: 1) durable remission profile (defined by the absence of thrombocytopenia, renal failure or clinical worsening for at least 30 days after the first day of normalisation of platelet levels), 2) refractory profile (defined by a platelet level after 4 days of intensive treatment of less than twice the initial level, associated with a persistently high level of lactate dehydrogenase), 3) relapse profile (defined by the recurrence of neurological manifestations, renal failure and/or thrombocytopenia < 100,000/mm3 for at least 2 days without any other cause identified after durable remission). The prognosis for TTP remains burdened by a mortality rate of around 10% and a relapse rate of 40-50%. The cellular players in the pathogenic process, responsible for the production of autoantibodies in this particularly severe disease, are still poorly characterised. This high-affinity memory B lymphocyte response requires cooperation with T lymphocyte players, namely follicular helper T lymphocytes. The involvement of these specific lymphocyte populations has been highlighted in the literature on other autoimmune diseases mediated by pathogenic autoantibodies, but has been little studied in TTP. The current high mortality rate in TTP suggests that a better understanding of immunopathological processes is required. Based on the model of other autoimmune diseases, this project should make it possible to identify the presence, at diagnosis, of circulating memory B lymphocytes specific for ADAMTS13, and also circulating autoreactive follicular helper T lymphocytes. After treatment with rituximab, depletion of circulating ADAMTS13-specific memory B lymphocytes is expected.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* patients with TTP at any stage of diagnosis (acute phase, lasting remission or not, relapse)
* patients undergoing internal medicine at Rouen University Hospital
* people who have read and understood the information letter
* membership of a social security scheme

Exclusion Criteria:

- a person deprived of liberty by an administrative or judicial decision or a person placed under court protection/guardianship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with thrombotic thrombocytopenic purpura, whatever the stage of diagnosis (acute phase, lasting remission or not, relapse)
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2027-05-11 (Estimated)

PRIMARY OUTCOMES:
Identifying the presence of circulating autoreactive T lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Identifying the presence of circulating autoreactive T lymphocytes in patients with TTP using the ELISPOT technique (Demonstration of spots indicating the presence of gamma interferon-producing T lymphocytes)
Identify the presence of circulating autoreactive B lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Identifying the presence of circulating autoreactive B lymphocytes in patients with TTP using the ELISPOT technique (Demonstration of IL-21 spots and specific B lymphocytes producing anti-ADAMTS13 antibodies in response to the ADAMTS13 antigen)

SECONDARY OUTCOMES:
Study quantitative variations in circulating autoreactive T lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Study quantitative variations in circulating autoreactive T lymphocytes in patients with TTP (Definition Number of T lymphocytes producing gamma interferon and IL-21 in response to ADAMTS13 antigen as determined by ELISPOT)
Study quantitative variations in circulating autoreactive B lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Study quantitative variations in circulating autoreactive B lymphocytes in patients with TTP (define the number of specific B lymphocytes producing anti-ADAMTS13 antibodies as determined by ELISPOT)
Determine the phenotypic characteristics of circulating autoreactive T lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Determine the phenotypic characteristics of circulating autoreactive T lymphocytes in patients with TTP (Determination of the number of effector and memory T lymphocyte subpopulations specific for ADAMTS13 by ELISPOT)
Determine the phenotypic characteristics of circulating autoreactive B lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Determine the phenotypic characteristics of circulating autoreactive B lymphocytes in patients with TTP (Assessment of the number of mature B lymphocyte subpopulations that are naive or memory ADAMTS13 specific)
Quantitative variations in circulating autoreactive T lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Study quantitative variations in circulating autoreactive T lymphocytes according to the different evolutionary profiles of patients (Evaluation of the number of T lymphocytes producing gamma interferon and IL-21 in response to the ADAMTS13 antigen as determined by ELISPOT)
Quantitative variations in circulating autoreactive B lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Study quantitative variations in circulating autoreactive B lymphocytes according to the different evolutionary profiles of patients (Evaluate the number of specific B lymphocytes producing anti-ADAMTS13 antibodies as determined by ELISPOT)
Determine the phenotypic characteristics of circulating autoreactive T lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Determine the phenotypic characteristics of circulating autoreactive T lymphocytes in patients with TTP (Determination of the proportion of effector and memory T lymphocyte subpopulations specific for ADAMTS13 by ELISPOT)
Determine the phenotypic characteristics of circulating autoreactive B lymphocytes | At enrollment visit, Month 3, Month 6 and month 12
  Determine the phenotypic characteristics of circulating autoreactive B lymphocytes in patients with TTP (Assessment of the proportion of mature B lymphocyte subpopulations that are naive or memory ADAMTS13 specific)

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital,, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.